CLINICAL TRIAL: NCT00989677
Title: Rheumatoid Arthritis Disease Activity Monitor
Acronym: RADAM
Status: Completed | Type: Observational
Sponsor: Maxima Medical Center (Other)
Collaborators: Philips Research Europe (Unknown)
Responsible Party: R.N.J. de Nijs MD, Maxima Medical Centre
Other Study IDs: NL2568201508; Protocol 5014-080820
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis

SUMMARY:
Background of the study:

Rheumatoid Arthritis (RA) is an autoimmune disease. There are four stages of the disease:

1. Synovial inflammation
2. Swelling of synovium
3. Pannus formation
4. Advanced bone and cartilage destruction Currently, there is no cure for RA, making the disease a chronic condition. RA is more prevalent in elderly and women. With medication it is possible to delay the onset of complications. Over the last decade, the treatment of RA has changed. Where treatment was palliative until pain medication was ineffective, the treatment is now more aggressive with early administration of disease modifying drugs (DMARDs).

The treatment for RA is staged. First, the patient receives generic, low-cost drugs. If this treatment becomes ineffective, the treatment is adjusted with different and usually more advanced drugs. Biologics are a category drugs that are considered most advanced and most expensive.

For effective treatment, there are two unmet needs.

* A tool to aid early diagnosis, as this allows early treatment and delay of complications and physical restrictions for patients.
* A safe, simple and cheap tool to monitor disease progress to allow traceable, operator-independent informed decisions on treatment adjustments.

Non-invasive optical methods offer several advantages over existing modalities. Optical contrast can be related to physiological parameters in the body, such as blood concentration and oxygenation. At relevant wavelengths and intensities, optical radiation is completely harmless. The cost of optical methods is low compared to other modalities. An important application, where optical methods can help diagnosis and treatment is detection of inflammation of joints in patients suffering from rheumatoid arthritis (RA). Due to the highly scattering nature of tissue, non-invasive optical methods for medical imaging are limited to the extremities of the human body. For application in joint diseases, this is acceptable, because imaging of hands can provide sufficient clinical information.

Objective of the study:

Primary objectives:

This is a retrospective, nonrandomized controlled observational study, conducted in a single center to evaluate the potential of optical attenuation measurements to establish disease activity for rheumatoid arthritis patients.

Secondary objectives:

Establish parameters from transient optical transmission measurements of the joint that relate to clinical evaluation results of individual joints Evaluate relation between disease activity (DAS-28 score) and the optical attenuation spectra of the fingers of a patient.

Study design:

This is a cross sectional, nonrandomized controlled observational study, conducted in a single center to evaluate the potential of optical attenuation measurements to establish disease activity for rheumatoid arthritis patients.

Study population:

The subject population will be patients visiting the Regionaal Reuma Centrum Eindhoven for rheumatoid arthritis. Patient visiting this center will represent a cross section of RA patients that are taken care of in an outpatient setting.

Primary study parameters/outcome of the study:

Primary endpoint is a successful measurement of optical attenuation of a joint and the part of the finger next to the joint before, during and after two consecutive restrictions of venous blood flow by means of a pressure cuff.

Secondary study parameters/outcome of the study (if applicable):

Secondary endpoints are unsuccessful measurements related to early termination of the measurement related to patient discomfort or safety and equipment or software failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Rheumatoid Arthritis
* Inflamed PIP joint of at least one index finger (moderate or severe)
* Disease activity of specific joints known (swelling, tenderness)
* No significant deformations of the hand or fingers
* More than 18 years old

Exclusion Criteria:

* Recent surgery or operation, in the last three months, on the arm or fingers that will be tested with the RADAM RRC
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will be patients visiting the Regionaal Reuma Centrum Eindhoven for rheumatoid arthritis. Patient visiting this center will represent a cross section of RA patients that are taken care of in an outpatient setting.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is a successful measurement of optical attenuation of a joint and the part of the finger next to the joint before, during and after two consecutive restrictions of venous blood flow by means of a pressure cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Ron NJ de Nijs, MD, Principal Investigator — Maxima Medical Center
Locations (1):
- Maxima Medical Centre, Eindhoven, Netherlands